CLINICAL TRIAL: NCT06059209
Title: The Role of Milk Fat Globule Membrane and 2'-Fucosyllactose in the Infant Gut Microbiota
Brief Title: Enfamil NeuroPro Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00000917
Record Dates: First submitted 2023-08-30; First posted 2023-09-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Infant Development; Infant ALL
Keywords: Healthy Infants

STUDY DESIGN:
Intervention Model Description: Subjects will be able to choose between the breast-fed or formula-fed group. Subjects in the formula-fed group will be randomly assigned to one of the two formulas, with a 50% chance of being assigned to each group.
Who Masked: Participant
Masking Description: Participants and research nurse/coordinator will be blinded to the formula assignment. The formulas used will be a standard infant formula (Enfamil Infant) and a new infant formula designed to be more similar to breast milk (Enfamil NeuroPro); both formulas are available for purchase by the public and meet FDA requirements for infant formulas. Each formula can (identical size) will be relabeled and coded by the investigators. Participants in the formula group will be provided with a four-month supply of powdered formula at the time of discharge from the hospital, along with stool collection kits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breast Milk (No Intervention)
- Enfamil Infant (Other)
  Interventions: Dietary Supplement: Enfamil Infant
- Enfamil NeuroPro (Active Comparator)
  Interventions: Dietary Supplement: Enfamil NeuroPro

INTERVENTIONS:
Dietary Supplement: Enfamil NeuroPro — FDA Infant formula
  Arms: Enfamil NeuroPro
Dietary Supplement: Enfamil Infant — FDA Infant formula
  Arms: Enfamil Infant

SUMMARY:
This study will compare infant gut bacteria for infants who have been fed a standard infant formula (Enfamil Infant); infants who have been fed a new infant formula designed to be more similar to breast milk (Enfamil NeuroPro); and breastfed infants. These formulas are currently available on the market and meet FDA requirements for infant formula.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, parallel-group study comparing breast milk to Enfamil Infant and Enfamil NeuroPro formulas. The central hypothesis of the study is that the addition of milk fat globule membrane and2'-Fucosyllactose (2'-FL) to infant formula plays a role in shaping the microbiota in a manner similar to the microbiota of breastfed infants. To test this hypothesis, the investigators will explore longitudinal changes in the fecal microbiome from birth to 4 months of age in infants fed breast-milk, standard Enfamil Infant formula or Enfamil NeuroPro formula. Fecal samples will be collected at birth, and then monthly for 4 months. At the time of last collection one serum sample will be collected. The investigators will analyze basic growth parameters, fecal microbial community analysis by metagenomics, fecal metabolome by untargeted metabolomic analysis, and fecal and systemic indicators of inflammation and intestinal barrier function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants with parental consent
* Parents are able to provide informed consent; own a smart phone and are able to fill out weekly digital questionnaires.

Exclusion Criteria:

* Prematurity (<= 36 weeks gestational age)
* Babies born through c-section
* Any health issues identified at the first postpartum screening
* Use of both breast milk and formula
* Use of donor breast milk
* Parent unwillingness/inability to avoid giving prebiotics, probiotics, symbiotics, and immune-stimulating products to the child for the duration of this study

Ages: 0 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in microbial DNA in term infants fed Enfamil NeuroPro as compared to standard Enfamil Infant formula or breast milk. | Birth to 4 months
  Assessed using 16S amplicon profiling of stool samples
Change from baseline in the gut metagenomics in term infants fed Enfamil NeuroPro as compared to standard Enfamil Infant formula or breast milk. | Birth to 4 months
  Samples sequenced using the NextSeq 500/550 and mapped against functional reference sequence databases using Bowtie2
Change from baseline of metabolome in term infants fed Enfamil NeuroPro as compared to standard Enfamil Infant formula or breast milk. | Birth to 4 months
  Untargeted analysis by automated comparison of the ion features in the experimental samples to a reference library of chemical standard entries.

SECONDARY OUTCOMES:
Growth- Height | Birth to 4 months
  Measured periodically in centimeters as part of routine care
Growth- Head circumference | Birth to 4 months
  Measured periodically in centimeters as part of routine care
Growth- Weight | Birth to 4 months
  Measured periodically in kg as part of routine care

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Data and specimens will not be stored for future research.